CLINICAL TRIAL: NCT03492307
Title: Weight-based Flow Rates for Children With Bronchiolitis on High-Flow Nasal Cannula: A Pilot Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: South Shore Hospital (Other)
Responsible Party: Principal Investigator, Alla Smith, Principal Investigator, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00028533
Record Dates: First submitted 2018-04-03; First posted 2018-04-10 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Bronchiolitis
Keywords: High Flow Nasal Cannula
MeSH Terms: conditions — Bronchiolitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Flow Protocol (Active Comparator): Patients randomized to this arm will receive HFNC according to our current protocol with a maximum of 8L/min.
  Interventions: Other: Standard Flow for HFNC (Maximum 8L/minute)
- Weight-Based Flow Protocol (Experimental): Patients randomized to this arm will receive HFNC according to a weight-based algorithm at 2L/kg/min.
  Interventions: Other: Weight-Based Flow for High Flow Nasal Cannula (HFNC) (2L/kg/minute)

INTERVENTIONS:
Other: Weight-Based Flow for High Flow Nasal Cannula (HFNC) (2L/kg/minute) — A weight-based flow for HFNC.
  Arms: Weight-Based Flow Protocol
Other: Standard Flow for HFNC (Maximum 8L/minute) — Maximum flow of 8L/minute.
  Arms: Standard Flow Protocol

SUMMARY:
This is a pilot study comparing a weight-based high-flow nasal cannula (HFNC) protocol with the current standard HFNC protocol for children <2yo admitted to South Shore Hospital with bronchiolitis. We currently use a flat limit of 8 liters of HFNC to support work of breathing and hypoxia in these patients. We will compare that to a weight-based protocol, which will provide 2L/kg/min of flow (flows generally between 6 and 20L/minute) to this patient population. The goal of this pilot study is to assess the feasibility of our study design. We will evaluate the functionality of a new weight-based flow protocol. We will also evaluate the functionality of a new bronchiolitis scoring tool, the Bronchiolitis Assessment Severity Score (BASS), and it's ability to guide care through the new protocol. We are also testing the feasibility of recruitment, randomization and retention. We are ultimately interested in whether a weight-based flow protocol reduces need for escalation to ICU-level care for children with moderate-severe bronchiolitis on HFNC.

DETAILED DESCRIPTION:
This is a pilot study comparing a weight-based high-flow nasal cannula (HFNC) protocol with the current standard HFNC protocol for children <2yo admitted to South Shore Hospital with bronchiolitis. We currently use a flat limit of 8 liters of HFNC to support work of breathing and hypoxia in these patients. We will compare that to a weight-based protocol, which will provide 2L/kg/min of flow (flows generally between 6 and 20L/minute) to this patient population. The goal of this pilot study is to assess the feasibility of our study design. We will evaluate the functionality of a new weight-based flow protocol. We will also evaluate the functionality of a new bronchiolitis scoring tool, the Bronchiolitis Assessment Severity Score (BASS), and it's ability to guide care through the new protocol. We are also testing the feasibility of recruitment, randomization and retention. We are ultimately interested in whether a weight-based flow protocol reduces need for escalation to ICU-level care for children with moderate-severe bronchiolitis on HFNC.

ELIGIBILITY:
Inclusion Criteria:

* admission to inpatient pediatrics
* clinical diagnosis of bronchiolitis
* BASS score of moderate or severe

Exclusion Criteria:

* non-english speakers
* patients with urgent need for CPAP, BIPAP or intubation

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Treatment failure | During hospital admission
  Need for escalation to NIV (CPAP or BIPAP) or intubation
Length of Stay | During hospital admission
  Length of hospital stay (admission to discharge or transfer)

CONTACTS AND LOCATIONS:
Overall Officials: Alla Smith, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- South Shore Hospital, Weymouth, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Smith A, Banville D, O'Rourke C, Melvin P, Batey L, Borgmann A, Waltzman M, Agus MSD. Randomized Trial of Weight-Based Versus Fixed Limit High-Flow Nasal Cannula in Bronchiolitis. Hosp Pediatr. 2023 May 1;13(5):387-393. doi: 10.1542/hpeds.2022-006656. PMID 37122050